CLINICAL TRIAL: NCT02791165
Title: Using Cardiac MRI to Characterise the Dynamic Changes Which Occur in the Acutely Reperfused STEMI Patient
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/3033
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-05

CONDITIONS: STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from all participants.
Oversight: Data Monitoring Committee: No

SUMMARY:
There is an optimal day on which to perform the CMR scan which allows one to capture the information required to assess the dynamic changes in the reperfused STEMI patient. The main objective is to characterise the dynamic changes in LV function, MI size, myocardial edema, MVO, IMH, interstitial volume in the remote myocardium over the first 10 days of an acute reperfused STEMI in order to identify the optimal day for performing the CMR scan.

DETAILED DESCRIPTION:
This will be a prospective observational study with serial CMR imaging only.

CMR scan Each patient will receive one CMR scan performed on Day 1, Day 3, Day 5, Day 10 following the PPCI procedure on a 3T Philips scanner (see study flow below). All CMR scans will be analysed at a central CMR corelab.

For Day 1, 3, 5, 7 and 10 CMRs, parameters will be collected as follows:

* Left ventricle (LV) ejection fraction and indexed LV end systolic and diastolic volumes and mass using short-axis SSFP cine imaging and myocardial tagging sequences).
* The AAR by T1 and T2 mapping18 as a percentage of the LV over time.
* Signal intensity of T1 and T2 mapping in the MI zone, MI core and remote myocardium over time.
* The incidence of intramyocardial haemorrhage (IMH)(hypo-enhancement on T2* mapping sequence)26.
* The volume of microvascular obstruction (MVO) defined as signal intensity 2 standard deviated below the mean signal intensity of the remote myocardium on the T2* maps.

Additional sequence for Day 3 and 7 CMR scans:

• All the above plus MI size (measured in mass of LGE and expressed as a percentage of the LV mass).

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed STEMI as per PPCI procedure reports/ clinical notes
2. Proximal to mid coronary artery occlusion.
3. Ability to provide informed consent

Exclusion Criteria:

1. Previous myocardial infarction or coronary artery bypass graft surgery
2. Contraindication for CMR (e.g. ferromagnetic implants, claustrophobia, estimated glomerular filtration rate <30mL/min)

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with an acute STEMI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | One year

CONTACTS AND LOCATIONS:
Overall Officials: National Heart Centre Singapore, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No